CLINICAL TRIAL: NCT00001685
Title: Immunization of HLA-A201 Patients With Metastatic Melanoma Using a Combination of Immunodominant Peptides From Three Melanoma Antigens, MART-1, GP100 and Tyrosinase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980023; 98-C-0023
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Cancer; IL-12; IL-2; Immunotherapy; Vaccine
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Neoplasms | interventions — MART-1 Antigen; Monophenol Monooxygenase

INTERVENTIONS:
Biological: Immunodominant peptides from three melanoma antigens, MART-1, GP100 and tyrosinase

SUMMARY:
This is a study of a melanoma tumor antigen peptide vaccine. Peptides representing HLA-A201 restricted T cell epitopes of the melanoma antigens, MART-1, gp100 and tyrosinase will be administered emulsified in Incomplete Freund's Adjuvant, (IFA) to HLA-A201 patients with melanoma. The study is designed to evaluate the potential therapeutic role, immunologic effects and toxicity of repeated doses of this peptide vaccine administered subcutaneously.

Immune reactivity to the peptide epitope will be monitored in all patients by analysis of melanoma-specific T cell precursors prior to and after immunization.

DETAILED DESCRIPTION:
This is a study of a melanoma tumor antigen peptide vaccine. Peptides representing HLA-A201 restricted T cell epitopes of the melanoma antigens, MART-1, gp100 and tyrosinase will be administered emulsified in Incomplete Freund's Adjuvant, (IFA) to HLA-A201 patients with melanoma. The study is designed to evaluate the potential therapeutic role, immunologic effects and toxicity of repeated doses of this peptide vaccine administered subcutaneously.

Immune reactivity to the peptide epitope will be monitored in all patients by analysis of melanoma-specific T cell precursors prior to and after immunization.

ELIGIBILITY:
Any patient 16 years of age or older with measurable metastatic melanoma who has failed standard treatment and has an expected survival of greater than three months.

Must be HLA-A0201.

Serum creatinine of 2.0 mg/dl or less.

Bilirubin 1.6 mg/dl or less.

WBC 3000/mm(3) or greater.

Platelet count 90,000 mm(3) or greater.

Serum AST/ALT less then two times normal.

ECOG performance status of 0 or 1.

Patients of both genders must be willing to practice effective birth control during the trial.

Must not be undergoing or have undergone in the past 3 weeks any other form of therapy except surgery for their cancer.

Must not have active systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular or respiratory systems or any known immunodeficiency disease.

Must not require steroid therapy.

Must not be pregnant.

Must not be positive for hepatitis B(s)AG or HIV antibody.

Must not have had a known allergic reaction to Incomplete Freund's Adjuvant (IFA).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114
Dates: Start 1997-11; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA. Cancer vaccines based on the identification of genes encoding cancer regression antigens. Immunol Today. 1997 Apr;18(4):175-82. doi: 10.1016/s0167-5699(97)84664-6. No abstract available. PMID 9136454
- [Background] Rosenberg SA. Development of cancer immunotherapies based on identification of the genes encoding cancer regression antigens. J Natl Cancer Inst. 1996 Nov 20;88(22):1635-44. doi: 10.1093/jnci/88.22.1635. PMID 8931607
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Dudley ME, Schwarz SL, Spiess PJ, Wunderlich JR, Parkhurst MR, Kawakami Y, Seipp CA, Einhorn JH, White DE. Immunologic and therapeutic evaluation of a synthetic peptide vaccine for the treatment of patients with metastatic melanoma. Nat Med. 1998 Mar;4(3):321-7. doi: 10.1038/nm0398-321. PMID 9500606